CLINICAL TRIAL: NCT04613895
Title: A Multi-Center, Open-label, Randomized Trial to Evaluate the Efficacy and Safety Based on Timing of Administration of DWP14012 in Patients With Erosive Esophagitis
Brief Title: Treatment Effect According to Timing of Administration of DWP14012 40 mg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Collaborators: Hanyang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT_DWP14012001
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — fexuprazan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fed state group (Experimental): just after a meal
  Interventions: Drug: DWP14012
- fasted state group (Experimental): before a meal
  Interventions: Drug: DWP14012

INTERVENTIONS:
Drug: DWP14012 — DWP14012 40 mg, orally, once daily just after a meal up to 4 weeks
  Other Names: fed state
  Arms: fed state group
Drug: DWP14012 — DWP14012 40 mg, orally, once daily before a meal up to 4 weeks
  Other Names: fasted state
  Arms: fasted state group

SUMMARY:
The primary objective of this study is to establish noninferiority of efficacy of DWP14012 (40 mg once daily) based on Timing of Administration.

DETAILED DESCRIPTION:
Subjects will provide written informed consent for study participation and then undergo appropriate screening. Subjects who meet the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to either before meal group or after meal group. Subjects will be stratified into two groups according to Los Angeles classification grades (LA grades) A/B or C/D, as determined by upper gastrointestinal (GI) endoscopy. Subjects will visit the site at Week 2 for endoscopic assessment. Subjects whose mucosal breaks have completely healed will be prematurely withdrawn and considered to have reached end of treatment. Subjects whose mucosal breaks have not healed will continue to receive IPs for an additional 2 weeks and will visit the site for endoscopic assessment at Week 4.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 19 and 75 years old based on the date of written agreement
* Those who have been diagnosed with erosive esophagitis of LA Grade A-D on the upper gastrointestinal endoscopy
* Those who experienced symptoms of heartburn or acid regurgitation within the last 7 days

Exclusion Criteria:

* Those who have undergone gastric acid suppression or gastric, esophageal surgery
* Those who with clinically significant liver, kidney, nervous system, respiratory, endocrine, hematologic, cardiovascular, urinary system disease

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2020-11-17 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
healing rate at 4 week | 4 week
  Cumulative healing rate of erosive esophagitis at 4 week by endoscopy

SECONDARY OUTCOMES:
healing rate at 2 week | 2 week
  Cumulative healing rate of erosive esophagitis at 2 week by endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No